CLINICAL TRIAL: NCT03811418
Title: Phase III Study to Compare Trastuzumab-biosimilar (Kanjinti®) Plus Pertuzumab Plus Vinorelbine With Trastuzumab-biosimilar (Kanjinti®) Plus Pertuzumab Plus Docetaxel as First-line Treatment for HER2-positive Advanced Breast Cancer
Brief Title: A Study to Compare Pertuzumab + Trastuzumab + Vinorelbine vs. Placebo + Trastuzumab + Docetaxel in Previously Untreated HER2-positive Metastatic Breast Cancer
Acronym: ATTILA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study approved with treatment regimen based on current guidelines. However, reimbursement of IMP was not feasible.
Sponsor: iOMEDICO AG (Industry)
Collaborators: Arbeitsgemeinschaft fur Internistische Onkologie (Other); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: iOM-110383; 2017-004749-25 (EudraCT Number)
Record Dates: First submitted 2018-12-13; First posted 2019-01-22 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-04

CONDITIONS: Advanced Breast Cancer; HER2-positive Breast Cancer
Keywords: advanced breast cancer; HER2-positive; metastatic; inoperable; female; quality of life
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Trastuzumab; pertuzumab; Vinorelbine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kanjinti/Pertuzumab plus Vinorelbine (Experimental): Patients will receive Kanjinti® (trastuzumab-biosimilar) plus pertuzumab plus vinorelbine.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Vinorelbine
- Kanjinti/Pertuzumab plus Docetaxel (Active Comparator): Patients will receive Kanjinti® (trastuzumab-biosimilar) plus pertuzumab plus docetaxel.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Trastuzumab — administered as combined therapy with pertuzumab and vinorelbine or docetaxel.
  Trastuzumab will be administered as an IV loading dose of 8 milligrams per kilogram (mg/kg) on day 1 of cycle 1 (1 cycle length = 21 days), and 6 mg/kg Q3W on day 1 of subsequent cycles until progressive disease, intolerable toxicity, or death.
  Other Names: Kanjinti®; ABP 980
Drug: Pertuzumab — administered as combined therapy with Kanjinti® and vinorelbine or docetaxel.
  Pertuzumab will be administered as an IV loading dose of 840 milligrams (mg) on day 1 of cycle 1 (1 cycle length = 21 days), and 420 mg Q3W on day 1 of subsequent cycles until progressive disease, intolerable toxicity, or death.
  Other Names: Perjeta®
Drug: Vinorelbine — administered as combined therapy with Kanjinti® and pertuzumab.
  Vinorelbine will be administered as an IV dose of 25 milligrams per kilogram (mg/kg) on days 1 and 8 of cycle 1 (1 cycle length = 21 days), and 25mg/kg up to 30 mg/kg (as per treating physician discretion) Q3W on day 1 of subsequent cycles until progressive disease, intolerable toxicity, or death.
  Arms: Kanjinti/Pertuzumab plus Vinorelbine
Drug: Docetaxel — administered as combined therapy with Kanjinti® and pertuzumab.
  Docetaxel will be administered as an IV dose of 75 milligrams per square meter (mg/m^2) on day 1 of cycle 1 (1 cycle length = 21 days), and 75 mg/m^2 (up to 100 mg/m^2 as per treating physician discretion) Q3W on day 1 of subsequent cycles until progressive disease, intolerable toxicity, or death.
  Arms: Kanjinti/Pertuzumab plus Docetaxel

SUMMARY:
This is a randomized, open-label, two-arm, phase III trial in Germany to investigate whether vinorelbine-based triple combination presents a less toxic treatment option than docetaxel-based triple combination in patients with HER2-positive advanced breast cancer who have not previously received any systemic treatment in the metastatic setting.

The primary objective of the study is to compare patient-reported quality of life in the two treatment arms. Patients will be followed-up for survival until death or end of study after at least 79 deaths occured in each arm, whatever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent prior to beginning of protocol-specific procedures.
* Histologically or cytologically confirmed adenocarcinoma of the breast. Locally advanced and inoperable or metastatic disease.
* HER2-positive disease, defined as IHC status HER2+++ or CISH/FISH status positive.
* Female patients aged ≥ 18 years.
* In case of adjuvant treatment, disease-free interval of at least 12 months after completion of adjuvant treatment (excluding hormonal therapy).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
* For women with childbearing potential, defined as physiologically capable of becoming pregnant:

  * Negative pregnancy test.
  * Agreement to use an effective form of contraception during study treatment and for 7 months after the last dose of study treatment.
* Life expectancy of at least 12 weeks.
* Adequate organ and bone marrow function
* Fluent in spoken and written German and willing to answer the questionnaires

Exclusion Criteria:

* Previous systemic treatment in palliative intention (chemotherapy, hormonal therapy and / or biological therapy)
* Persistent peripheral sensory or motor neuropathy grade 2 or higher (NCI CTCAE v5.0)
* Evidence of central nervous system metastases. CT or MRI of the brain is only mandatory in case of clinical suspicion of brain metastases
* Current uncontrolled hypertension (systolic > 150 mmHg and / or diastolic > 100 mmHg) or clinically significant cardiovascular disease
* History of LVEF < 50% during or after prior (neo)adjuvant therapy with trastuzumab
* Current severe, uncontrolled systemic disease (e.g. cardiovascular, pulmonary, or metabolic disease, wound healing disorder, ulcers, or bone fractures, or severe fungal, bacterial or viral infection)
* Major surgery within 28 days prior to start of study medication, or anticipation of the need for major surgery during the course of study treatment
* Current known infection with HIV, HBV, or HCV (testing not required)
* Dyspnea at rest due to complications of advanced malignancy, or other diseases requiring continuous oxygen therapy.
* Known hypersensitivity to any of the study medications or to excipients of recombinant human or humanized antibodies.
* Participation in investigational studies within 30 days or five half-lives of the respective IMP, whichever is longer, prior randomization.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Patient-reported health-related quality of life (QoL): FACT-B | Baseline to week 18
  Area under the curve (AUC) in the Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire subscale Trial Outcome Index-Physical/Functional/Breast (TOI-PFB) after 18 weeks (irrespective of disease or treatment situation at that time point). Higher AUC indicates better quality of life.
  To calculate the TOI-PFB the three subscales Physical well-being (PWB - 7 statements), Functional well-being (FWB - 7 statements) and breast cancer subscale (BCS - 10 statements) are summed up. In all subscales each statement will be rated by the patient from 0 (not at all) - 4 (very much). Therefore ranges of subscales are: PWB 0 - 28; FWB 0 - 28; BCS 0 - 40; TOI-PFB 0 - 96; higher values indicate better quality of life.

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed by the investigator | Baseline, every 12 weeks after randomization (maximum up to 76 months)
  PFS is defined as time from randomization to date of progressive disease or death, whichever comes first. It will be analyzed using Kaplan-Meier method. Data will be censored at date of last contact for patients alive without progressive disease at database lock. If subsequent treatment was started prior to progressive disease, then data will be censored at the onset of this treatment.
Overall survival (OS) | Time from randomization to date of death (maximum up to approximately 76 months)
  OS is defined as time from randomization to date of death. It will be analyzed using Kaplan-Meier method. Data will be censored at date of last contact for patients alive at database cut/lock.
Overall response rate (ORR) | Baseline, every 12 weeks after randomization (maximum up to 76 months)
  Overall response rate is defined as the proportion of patients achieving a complete or partial remission as best response.
Clinical benefit rate (CBR) | Baseline, every 12 weeks after randomization (maximum up to 76 months)
  CBR is defined as proportion of patients achieving a complete or partial remission or a stable disease lasting at least 24 weeks.
Time to treatment failure (TTF) | Baseline, every 12 weeks after randomization (maximum up to 56 months)
  TTF is defined as time from randomization to discontinuation of all study medications. Date of discontinuation is the earliest end of last cycle (= 20 days after first administration of a study drug in the last cycle) OR progressive disease after last administration of any study drug OR death OR start of a subsequent treatment.
Incidence of (Serious) Adverse events ((S)AEs) | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  Type, frequency and severity of adverse events (including those from the pre- and post-treatment periods) will be listed according to Common Toxicity Criteria for Adverse Events (CTCAE).
Blood count: Hemoglobin | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  The amount of hemoglobin in the blood will be measured in g/dL as per clinical routine and will be displayed using by-patient listings.
Blood count: Platelet Count | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  The number of platelets in the blood will be counted as per clinical routine and will be displayed using by-patient listings.
Blood count: Leukocytes | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  The number of leukocytes in the blood will be counted as per clinical routine and will be displayed using by-patient listings.
Blood count: Absolute Neutrophil Count | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  The absolute neutrophil count will be determined as per clinical routine and will be displayed using by-patient listings.
Safety monitoring (coagulation): Coagulation (INR) | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  Coagulation (INR) as per clinical routine will be displayed using by-patient listings.
Clinical chemistry: Alkaline Phosphatase | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  Alkaline phosphatase will be measured in U/L as per clinical routine and will be displayed using by-patient listings.
Clinical chemistry: Alanine transaminase (ALT) | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  ALT will be measured in U/L as per clinical routine and will be displayed using by-patient listings.
Clinical chemistry: Aspartate transaminase (AST) | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  AST will be measured in U/L as per clinical routine and will be displayed using by-patient listings.
Clinical chemistry: Bilirubin total | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  Total bilirubin will be measured in mg/dL as per clinical routine and will be displayed using by-patient listings.
Clinical chemistry: Creatinine (Serum) | From date of informed consent to +30 days from last application of study medication (maximum up to 57 months)
  Serum creatinine will be measured in µmol/L as per clinical routine and will be displayed using by-patient listings.
Left Ventricular Ejection Fraction (LVEF) monitoring | LVEF at baseline, every three months thereafter until end of treatment, then every six months for 24 months thereafter (maximum up to 76 months)
  Incidence of clinically relevant LVEF levels. Change from baseline at each assessment time point, worst-on-treatment will be displayed using descriptive statistics.
Patient-reported health-related quality of life (QoL): Trial Outcome Index-Physical/Functional/Breast (TOI-PFB) | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  AUC in TOI-PFB at 12, 18, 24 and 36 months.
  Area under the curve (AUC) in the Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire subscale Trial Outcome Index-Physical/Functional/Breast (TOI-PFB) after 12, 18, 24 and 36 months (irrespective of disease or treatment situation at that time point). Higher AUC indicates better quality of life.
  To calculate the TOI-PFB the three subscales Physical well-being (PWB - 7 statements), Functional well-being (FWB - 7 statements) and breast cancer subscale (BCS - 10 statements) are summed up. In all subscales each statement will be rated by the patient from 0 (not at all) - 4 (very much). Therefore ranges of subscales are: PWB 0 - 28; FWB 0 - 28; BCS 0 - 40; TOI-PFB 0 - 96; higher values indicate better quality of life.
Patient-reported health-related quality of life (QoL): FACT-B TOI-PFB | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  Time to decline by 5 points in the Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire subscale Trial Outcome Index-Physical/Functional/Breast (TOI-PFB).
  To calculate the TOI-PFB the three subscales Physical well-being (PWB - 7 statements), Functional well-being (FWB - 7 statements) and breast cancer subscale (BCS - 10 statements) are summed up. In all subscales each statement will be rated by the patient from 0 (not at all) - 4 (very much). Therefore ranges of subscales are: PWB 0 - 28; FWB 0 - 28; BCS 0 - 40; TOI-PFB 0 - 96; decline of scale indicates worsening quality of life.
Patient-reported health-related quality of life (QoL): FACT-B total score | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  Change from baseline in the FACT-B total score for all questionnaire timepoints. To calculate FACT-B total score patient ratings from 0 (not at all) - 4 (very much) to each of the 37 questionnaire statement are summed up. Total score range: 0 - 148. Higher values indicate better quality of life
Patient-reported health-related quality of life (QoL): FACT-B subscale physical well-being (PWB) | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  Change from baseline in the FACT-B subscale PWB for all questionnaire timepoints. PWB subscale consists of 7 statements leading to a scale range of 0-28. Higher values indicate better quality of life
Patient-reported health-related quality of life (QoL): FACT-B subscale social/family well-being (SWB) | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  Change from baseline in the FACT-B subscale SWB for all questionnaire timepoints. SWB subscale consists of 8 statements leading to a scale range of 0-32. Higher values indicate better quality of life
Patient-reported health-related quality of life (QoL): FACT-B subscale emotional well-being (EWB) | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  Change from baseline in the FACT-B subscale EWB for all questionnaire timepoints. EWB subscale consists of 6 statements leading to a scale range of 0-24. Higher values indicate better quality of life
Patient-reported health-related quality of life (QoL): FACT-B subscale functional well-being (FWB) | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  Change from baseline in the FACT-B subscale FWB for all questionnaire timepoints. FWB subscale consists of 7 statements leading to a scale range of 0-28. Higher values indicate better quality of life
Patient-reported health-related quality of life (QoL): FACT-B breast cancer subscale (BCS) | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  Change from baseline in the FACT-B BCS score for all questionnaire timepoints. BCS consists of 10 statements leading to a score range of 0-40. Higher values indicate better quality of life
Patient-reported health-related quality of life (QoL): FACT-B breast cancer subscale (BCS) score decline | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  Time to decline by 2 points in the FACT-B BCS score. BCS consists of 10 statements leading to a score range of 0-40. BCS score decline indicates worsening quality of life.
Patient-reported health-related quality of life (QoL): FACT/GOG-Ntx4 subscale | Baseline, every three weeks for the first 24 weeks, every three months thereafter (maximum up to 36 months).
  Change from baseline in the FACT/GOG-Ntx4 subscale for all questionnaire timepoints. FACT/GOG-Ntx4 subscale consists of 11 statements leading to a scale range of 0-44. Higher values indicate better quality of life
Exploratory endpoint: Treatment costs | From randomization until end of treatment (maximum up to 56 months).
  Treatment costs (drug costs)
Exploratory endpoints: Duration of hospitalizations | From randomization until end of treatment (maximum up to 57 months).
  Total duration of hospitalizations (per patients)
Exploratory endpoints: Number of hospitalizations | From randomization until end of treatment (maximum up to 57 months).
  Number of hospitalizations (in-patient stays)
Exploratory endpoints: Reasons for hospitalizations | From randomization until end of treatment (maximum up to 57 months).
  Reasons for hospitalizations
Exploratory endpoints: Febrile infections | From randomization until end of treatment (maximum up to 57 months).
  Incidence of febrile infections
Exploratory endpoints: Employment status | From randomization until end of treatment (maximum up to 56 months).
  Employment status (kind and duration of sick leaves)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Welt, Dr., Principal Investigator — Essen University Hospital
Locations (1):
- iOMEDICO AG, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson M, Lidbrink E, Bjerre K, Wist E, Enevoldsen K, Jensen AB, Karlsson P, Tange UB, Sorensen PG, Moller S, Bergh J, Langkjer ST. Phase III randomized study comparing docetaxel plus trastuzumab with vinorelbine plus trastuzumab as first-line therapy of metastatic or locally advanced human epidermal growth factor receptor 2-positive breast cancer: the HERNATA study. J Clin Oncol. 2011 Jan 20;29(3):264-71. doi: 10.1200/JCO.2010.30.8213. Epub 2010 Dec 13. PMID 21149659
- [Background] Andersson M, Lopez-Vega JM, Petit T, Zamagni C, Easton V, Kamber J, Restuccia E, Perez EA. Efficacy and Safety of Pertuzumab and Trastuzumab Administered in a Single Infusion Bag, Followed by Vinorelbine: VELVET Cohort 2 Final Results. Oncologist. 2017 Oct;22(10):1160-1168. doi: 10.1634/theoncologist.2017-0079. Epub 2017 Jun 7. PMID 28592618
- [Background] Baselga J, Cortes J, Kim SB, Im SA, Hegg R, Im YH, Roman L, Pedrini JL, Pienkowski T, Knott A, Clark E, Benyunes MC, Ross G, Swain SM; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med. 2012 Jan 12;366(2):109-19. doi: 10.1056/NEJMoa1113216. Epub 2011 Dec 7. PMID 22149875
- [Background] Burstein HJ, Keshaviah A, Baron AD, Hart RD, Lambert-Falls R, Marcom PK, Gelman R, Winer EP. Trastuzumab plus vinorelbine or taxane chemotherapy for HER2-overexpressing metastatic breast cancer: the trastuzumab and vinorelbine or taxane study. Cancer. 2007 Sep 1;110(5):965-72. doi: 10.1002/cncr.22885. PMID 17614302
- [Background] Cortes J, Baselga J, Im YH, Im SA, Pivot X, Ross G, Clark E, Knott A, Swain SM. Health-related quality-of-life assessment in CLEOPATRA, a phase III study combining pertuzumab with trastuzumab and docetaxel in metastatic breast cancer. Ann Oncol. 2013 Oct;24(10):2630-2635. doi: 10.1093/annonc/mdt274. Epub 2013 Jul 17. PMID 23868905
- [Background] Perez EA, Lopez-Vega JM, Petit T, Zamagni C, Easton V, Kamber J, Restuccia E, Andersson M. Safety and efficacy of vinorelbine in combination with pertuzumab and trastuzumab for first-line treatment of patients with HER2-positive locally advanced or metastatic breast cancer: VELVET Cohort 1 final results. Breast Cancer Res. 2016 Dec 13;18(1):126. doi: 10.1186/s13058-016-0773-6. PMID 27955684
- [Background] Swain SM, Baselga J, Kim SB, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Heeson S, Clark E, Ross G, Benyunes MC, Cortes J; CLEOPATRA Study Group. Pertuzumab, trastuzumab, and docetaxel in HER2-positive metastatic breast cancer. N Engl J Med. 2015 Feb 19;372(8):724-34. doi: 10.1056/NEJMoa1413513. PMID 25693012